CLINICAL TRIAL: NCT05821699
Title: Implementing and Evaluating the Effect of Personalized Pain Coaches After Orthopaedic Surgery for Patients With Sports Medicine Injuries to Improve Postoperative Outcomes
Brief Title: Effect of Personalized Pain Coaches After Orthopaedic Surgery for Patients With Sports Medicine Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Football League (Other)
Responsible Party: Principal Investigator, Nicholas A. Giordano, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004925
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sports Medicine Injuries
Keywords: Personalized Pain Coach; Postoperative outcome; Life Care Specialist
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In Person LCS Intervention- With Opioid Risk Education (Experimental): Patients will receive opioid education and Naloxone education. Therapeutic Intervention will include education on implementing mindfulness practices into postoperative recovery, known as the Community Resiliency Model CRM). Clinical Pain Coordination will include directed referrals for complex needs, including mental health and substance use disorders, as needed. All participants in the LCS intervention arm will also receive the current standard-of-care. The Community Resiliency Model (CRM) is a noncognitive variant of mindfulness, emphasizing attunement to interoceptive and exteroceptive signaling cues for regulation of autonomic responses to stress. CRM skills are introduced over a sixty-to-ninety-minute session, allowing for a brief introduction and application of skills by participants. These will be in person.
  Interventions: Behavioral: LCS (Life Care Specialist)
- Virtual LCS Intervention-With Opioid Risk Education (Experimental): Participants will receive opioid education, and Naloxone education. Therapeutic Intervention will include education on implementing mindfulness practices into postoperative recovery, known as the Community Resiliency Model CRM). Clinical Pain Coordination will include directed referrals for complex needs, including mental health and substance use disorders, as needed. All participants in the LCS intervention arm will also receive the current standard-of-care. The Community Resiliency Model (CRM) is a noncognitive variant of mindfulness, emphasizing attunement to interoceptive and exteroceptive signaling cues for regulation of autonomic responses to stress. CRM skills are introduced over a sixty-to-ninety-minute session, allowing for a brief introduction and application of skills by participants. These will be in performed virtually via a digital conferencing platform
  Interventions: Behavioral: LCS (Life Care Specialist)
- No LCS intervention (Active Comparator): Patients will receive the current standard-of-care for pain management in the aftermath of surgery, which includes: a standardized prescription protocol, hospital-system approved discharge instructions which provide written instruction on how to taper opioid use, links to written/online resources for opioid misuse, overdose prevention, and State-approved disposal options.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: LCS (Life Care Specialist) — The LCS will work with the patient to create a pain management plan focused on behavioral education. The LCS interventions can encompass all, but not limited to, the information included below:
  * Opioid Risk Education
  * Therapeutic Intervention
  * Clinical Pain Coordination
  Arms: In Person LCS Intervention- With Opioid Risk Education; Virtual LCS Intervention-With Opioid Risk Education
Behavioral: Standard of Care — Patients will receive the current standard-of-care for pain management in the aftermath of surgery: a standardized prescription protocol, hospital-system approved discharge instructions which provide written instruction on how to taper opioid use, links to written/online resources for opioid misuse, overdose prevention, and State-approved disposal options.
  Arms: No LCS intervention

SUMMARY:
Patients experiencing sports medicine-related injuries are particularly vulnerable to developing both chronic pain and experiencing prolonged opioid use. This multiarmed randomized controlled trial will quantify the impact of integrating Life Care Specialists, and pain management-focused paraprofessionals, have on increasing access to multimodal pain management approaches and subsequently optimizing both patient-reported pain-related outcomes and objective measures of activity. Life Care Specialists work with patients and clinicians on implementing non-pharmacological pain management approaches, specifically teaching participants how to implement mindfulness-based skills into their recovery, systematically conducting standardized biopsychosocial pain assessments, and coordinating care. By developing a toolbox of pain management approaches with the support of the Life Care Specialist, patients are well positioned to incorporate evidence-based pain management approaches into their recovery that result in improved psychosocial functioning and reduced opioid medication utilization. In total, 150 individuals with sports medicine injuries will be randomized to one of two intervention arms where they will work with a Life Care Specialist in person or over telehealth or receive standard-of-care written postoperative instructions for pain management. Patient-reported outcomes, objective actigraphy movement outcomes captured using wrist-based watches, and opioid utilization captured using medication event monitoring system (MEMS) caps will be evaluated over 3-months postoperatively for a total of 4 study visits.

DETAILED DESCRIPTION:
Longitudinal analyses indicate that both greater pain severity and duration precede poor functioning and prolonged opioid use. This finding suggests that optimizing pain management, soon after painful events, such as orthopaedic injury, is vital to reducing risks related to prolonged opioid use. However, opioid-dominant pain management, which remains the standard of care across many health systems and in orthopaedic surgery, elevates the risks for ineffective pain management and, subsequently, opioid dependency by only targeting a select number of pain receptors.

Multimodal analgesia, which combines analgesic drugs from different classes and employs analgesic techniques that target multiple pain-related receptors, is recommended in the treatment of acute postoperative pain because its synergistic effect maximizes pain relief at lower analgesic doses, thereby reducing the risk of adverse opioid-related effects and chronic pain.

The study team's interdisciplinary team has developed and tested a novel clinical care team role focused on optimizing pain management after surgery, known as a Life Care Specialist. Life Care Specialists provide patient-centered pain management care coordination, teach patients how to implement non-pharmacological pain management approaches, and deliver opioid safety-focused pain education, not only during acute hospitalization but also throughout postoperative recovery.

Life Care Specialists provide pain-focused care coordination for patients with complex needs after orthopedic injury, including communicating patient care needs and goals of care to clinical care team members (e.g. surgeons, acute pain service, physical therapy, nursing staff), connecting patients to yoga instructors, massage therapists, and engaging behavioral health consults to work with patients over time to improve biopsychosocial pain presentations.

For this trial, 150 individuals with sports medicine injuries will be randomized to one of two intervention arms where they will work with a Life Care Specialist in person or over telehealth or receive standard-of-care written postoperative instructions for pain management. Patient-reported outcomes, objective actigraphy movement outcomes captured using wrist-based watches, and opioid utilization captured using MEMS caps will be evaluated over 3-months postoperatively for a total of 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 15-45 years old
* Scheduled for orthopedic surgery due to sports medicine injuries (e.g., anterior cruciate ligament tears, meniscus injury, rotator cuff injury, etc.), who are actively employed or full-time athletes before injury

Exclusion Criteria:

* Individuals unable to provide consent
* Those undergoing revision procedures
* Individuals without access to an internet-connected device
* Individuals who are unemployed or retired at the time of injury will be ineligible.
* Individuals who are incarcerated or pregnant will not be eligible.
* Individuals unable to communicate in English will be excluded since all surveys are validated in English.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes Pain numerical rating scale (NRS) | 1 month pre-surgery, 2 weeks, 6 weeks, and 3 months post-surgery
  The NRS requires respondents to rate the intensity of their pain on a defined scale from 0, "no pain", to 10, 'the worst pain imaginable". The NRS is a commonly used pain assessment tool in both clinical practice and research. However, the NRS is a single static measure of pain and does not capture the biopsychosocial presentations of pain including physical functioning. Inpatient NRS, which is recorded by the clinical care team throughout each day, will be extracted from the electronic health record (EHR) by study staff upon participants' discharge from the hospital
Changes to Opioid utilization | 1 month pre-surgery, 2 weeks, 6 weeks, and 3 months post-surgery
  Inpatient and operating room opioid utilization will be extracted from the electronic health record (EHR) by study staff upon participants' discharge from the hospital. Opioid medication dosage will be transformed to morphine milligram equivalent (MME). MME will be averaged over the length-of-stay (LOS) for a daily dosage, known as MME/day. Additionally, the study team will review participants' EHR at each study time point up to 3-months to determine MME throughout postoperative recovery and rehabilitation and review medication in MEMS cap.

SECONDARY OUTCOMES:
Changes in Opioid Overdose Knowledge Scale (OOKS) | 1 month pre-surgery, 2 weeks, 6 weeks, and 3 months post-surgery
  Each participant will complete a questionnaire evaluating knowledge of signs and symptoms of opioid-involved overdose and details of naloxone utilization, if applicable. Higher scores indicating greater knowledge on how to identify and appropriately intervene during an overdose
Changes to PROMIS | 1 month pre-surgery, 2 weeks, 6 weeks, and 3 months post-surgery
  Sleep Disturbance, Physical Function, Pain Interference, Prescription Pain Medication Misuse. These PROMIS measures capture their respective domains of health. Respondents report their capabilities to perform each task or symptom burden on a Likert scale from 5, "without any difficulty", to 1, "unable to do". All items' raw scores are summed before being transformed into t-scores ranging from 0 to 100. Higher scores are better and indicate greater physical function, whereas higher scores on the other domains indicate worse symptom presentation.
Changes in Mindful Attention Awareness Scale (MAAS) | 1 month pre-surgery, 2 weeks, 6 weeks, and 3 months post-surgery
  The MAAS is a validated 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present
Changes to Actigraphy based sleep and activity data | 1 month pre-surgery, 2 weeks post-surgery
  Study participants will be given a wrist actigraphy device during their hospitalization and recovery until their 2-week follow-up appointment with the surgical team or until the watch battery loses its charge, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Giordano, PhD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in articles, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months after study completions and ending 24 months after study completion
Access Criteria: Investigators whose proposed use of the data has been approved by the Emory IRB and their institution's affiliated IRB and any necessary data use agreements overseen by Emory. Requests should be sent directly to the PI via email summarizing the purpose of utilizing the data.